CLINICAL TRIAL: NCT01822626
Title: Pediatrician-lead Motivational Counselling to Control BMI in Overweight Children: a RCT in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: reggioemilia2013
Record Dates: First submitted 2013-03-28; First posted 2013-04-02 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Overweight
Keywords: overweight; obesity; children; BMI; counseling; pediatrician
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- motivational counseling (Experimental)
  Interventions: Behavioral: motivational counseling
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: motivational counseling — A family pediatrician-lead counselling was offered to children assigned to the intervention group. The counselling program consisted of 5 motivational interviews based on Stages of Change Theory. Child and family always had to leave the meeting having agreed two objectives, one concerning food and one physical activity improvements, clearly defined and achievable. During each subsequent interview was assessed the degree of achievement of the objectives of the previous meeting. Based on the assessment the objective could be reinforced or redefined. After each change the objectives were recorded.
  Arms: motivational counseling

SUMMARY:
Obesity is one of the leading causes of morbidity and mortality in the industrialised world. Evidence is growing that early life nutrition can play a role in behavioural and cognitive problems in children and adolescents and is well documented that being overweight and obese during childhood can have short- and long-term physical and psycho-social health implications.

This is an individually randomised trial to evaluate the efficacy of a family pediatrician-lead counselling intervention in reducing the BMI of over-weight children aged 4-7 years old. As secondary objectives the investigators evaluate the effect of the counselling on dietary behaviours and physical activity.

The investigators targeted the intervention to overweight children, while obese children were referred to specialised care. The counselling targeted diet, physical activity, and sedentary behaviours.

ELIGIBILITY:
Inclusion Criteria:

* overweight children with BMI percentile between 85° and 94°
* 4-7 years old
* resident in Reggio Emilia Province
* assisted by the pediatrician at least for 12 months

Exclusion Criteria:

* metabolic pathologies and all pathologies related with obesity
* family in pre-contemplation stage

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 372 (Actual)
Dates: Start 2011-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
BMI variation from baseline | 12 months
  Difference between 12-month BMI score (weight/heigh2) and time-0 BMI score. Intervention average and control average BMI score are compared by Wilcoxon-Mann Whitney Test.

SECONDARY OUTCOMES:
Physical Activity behaviors variations | 12 months
  Physical activity: variation from baseline and 12-month questionnaire in weekly frequency of organized and spontaneous physical activity, variation from baseline and 12-month questionnaire in daily hours of television and computer.
Diatary behaviors variations | 12 month
  Dietary behaviors: variation from baseline and 12-month questionnaire of consumption of foods and drinks.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Maria Davoli, Principal Investigator — Primary Care Program, Local Health Authority of Reggio Emilia, Italy
Locations (1):
- Local Health Authority of Reggio Emilia, Reggio Emilia, Italy, Italy

REFERENCES:
- [Derived] Davoli AM, Broccoli S, Bonvicini L, Fabbri A, Ferrari E, D'Angelo S, Di Buono A, Montagna G, Panza C, Pinotti M, Romani G, Storani S, Tamelli M, Candela S, Giorgi Rossi P. Pediatrician-led motivational interviewing to treat overweight children: an RCT. Pediatrics. 2013 Nov;132(5):e1236-46. doi: 10.1542/peds.2013-1738. Epub 2013 Oct 21. PMID 24144717